CLINICAL TRIAL: NCT06030856
Title: A Pilot Randomized Controlled Trial to Assess a Model of Decentralised STI-Self Testing and Risk Self-Assessment Among Adolescent Girls and Young Women in South Africa to Trigger PrEP Re-start
Brief Title: PrEP Restart for Adolescent Girls and Young Women Using STI Self Testing and Assessment of Risk
Acronym: PALESA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wits RHI Research Centre Clinical Research Site (Other)
Collaborators: University of Alabama at Birmingham (Other); University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Thesla Palanee-Phillips, Director:Clinical Trials, Wits RHI Research Centre Clinical Research Site
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PALESA
Record Dates: First submitted 2023-08-24; First posted 2023-09-11 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: HIV Prevention
Keywords: Pre-Exposure Prophylaxis; HIV; Sexually Transmitted Infection (STI)
MeSH Terms: conditions — Sexually Transmitted Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- STI test kits for home use coupled with self-administered behavioural risk assessment (Experimental): The adolescent will receive STI test kits (NG, CT and TV) for home use coupled with self-administered behavioural risk assessment at the screening and enrolment visit.
  Interventions: Device: STI test kits (NG, CT and TV) for home use; Behavioral: Self Administered Behavioural Risk Assessment
- Self-administered behavioural risk assessment only (standard of care) (Active Comparator): The adolescent will receive a self-administered behavioural risk assessment at the screening and enrolment visit
  Interventions: Behavioral: Self Administered Behavioural Risk Assessment

INTERVENTIONS:
Device: STI test kits (NG, CT and TV) for home use — The adolescent randomized to the at-home STI testing arm will be provided with in-person instruction at enrollment and flyers (in English and isiZulu) with printed step-by-step instructions for kit use. Information will include details on how to store the kits, criteria for adequate specimen collection and preparation, how to run the test, and how to interpret the test results. Video-based instructions with accompanying text subtitles and audio options may also be provided for home use.
  Arms: STI test kits for home use coupled with self-administered behavioural risk assessment
Behavioral: Self Administered Behavioural Risk Assessment — Self Administered assessment to determine risk of HIV, STIs and pregnancy

SUMMARY:
This is a pilot randomized trial among 50 AGYW (aged ≥16≤18 years), who discontinued PrEP use within the past 6 months, assigned in a 1:1 ratio to receive: 1) STI self-test kits (Neisseria gonorrhoea (NG), Chlamydia trachomatis (CT) and Trichomonas vaginalis (TV)) with in-person instruction at enrolment and telephone/video-based instructions for home use coupled with self-administered behavioural risk assessment or 2) self-administered behavioural risk assessment only (standard of care). All participants will receive comprehensive sexual and reproductive health (SRH) services during their study visits including choice of family planning method initiation and support, and behavioural HIV/STI risk reduction counselling.

DETAILED DESCRIPTION:
The PALESA study aims to determine the feasibility of conducting a randomized controlled trial (RCT) to determine the impact of decentralized sexually transmitted infection (STI) point of care (POC) self-testing and risk self-assessment interventions to trigger pre-exposure prophylaxis (PrEP) re-start among adolescent girls and young women (AGYW) in South Africa at potential ongoing risk of re- acquiring STIs and HIV.

This overall study comprises two components that include a formative research study enrolling ~60 participants for qualitative in-depth interviews (IDIs) (this has been completed) and a prospective cohort study (Pilot randomized controlled trial - RCT) enrolling 50 AGYW with both clinical, diagnostic laboratory and nested qualitative methodologies.

The RCT seeks to establish the feasibility of conducting a randomized controlled trial among AGYW in South Africa to determine the impact of decentralized or at-home STI testing [(for Neisseria gonorrhea (NG), Chlamydia trachomatis (CT) and Trichomonas vaginalis (TV)] on restarting PrEP relative to a self-administered behavioural risk assessment. Additionally qualitative interviews will be conducted to assess adolescent girls experiences of at-home STI testing, behavioural risk assessment, and re-starting PrEP while participating in the pilot trial through exit interviews.

Objective 1: To determine the feasibility and acceptability of conducting a RCT among South African AGYW to determine the impact of STI self-testing coupled with a self-administered behavioural risk assessment on restarting PrEP relative to a self-administered behavioural risk assessment only

Objective 2: To assess AGYW acceptability of and experiences with use at-home STI testing, self-administered behavioural risk assessment, and re-starting PrEP while participating in the pilot RCT

ELIGIBILITY:
Inclusion Criteria:

* For the full cohort, all participants must:

  * Be cis-gender adolescent females (16-20 years of age)
  * Be literate
  * Currently sexually active
  * Be willing to participate in in-person and virtual study visits
  * Not be pregnant or planning to be pregnant for the next 6 months
  * Be HIV-negative but not ready to initiate PrEP at the screening and enrolment visit
  * Have used PrEP with subsequent discontinuation within the last 6 months
  * Have no contraindications to oral PrEP per self-report
  * Have no indication of possible acute HIV infection, according to South African PrEP guidelines
  * Have their own personal smart phone
  * Willing to provide written informed consent/assent to participate in this study

For the subset invited to qualitative interviews, all participants must be:

• Willing to participate in an IDI at/before their month 6 visit (study exit visit)

Exclusion Criteria:

* Potential AGYW participants who meet any of the following criteria will be excluded from the study:

  * At Screening and Enrollment, parent/guardian (for those participants <18 years) is unwilling to provide written informed consent
  * At Screening and Enrollment, is already participating in another research study involving drugs, medical devices, or vaccines for STI prevention or treatment.
  * Is not willing to comply with study procedures
  * As determined by the PIs/designee, any current or historical physical health, mental health or social issue or condition that the site investigator or designee determines should exclude participation.
  * Has any other condition that, in the opinion of the PIs/designee, would preclude informed consent, make study participation unsafe, or otherwise interfere with achieving the study objectives.

Ages: 16 Years to 20 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-07-05 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Number of participants enrolled and retained in the PALESA study | 1 year
  A recruitment target of 50 adolescent girls and young women and over 90% retention of those participants is achieved
Assessing Risk of Acquiring HIV and STIs | 1 year
  A self administered behavioural risk assessment questionnaire with 16 - 20 questions (which include questions on STI test results), which will tally up a score, will be used to measure how much counselling and guidance will the participants need to restart PrEP.
  A score of 0 - 7 means medium recommendation to restart PrEP. A score 8-15 means a strong recommendation to restart PrEP. Test results of STIs from the self-testing STI kit are shared on the self-administered behavioural risk assessment questionnaire.
Number of participants that restarted PrEP | 1 year
  There will be a dispensation form for every participant, this form will indicate if PrEP was restarted by the participant, and it will calculate include pill counts when PrEP bottles are returned to the research site
PrEP continuation 1 month after re-start | 1 year
  Dried Blood Spot (DBS) collected to measure tenofovir diphosphate (TFV-DP) level as an objective assessment of adherence to PrEP.
Experiences of at-home STI testing, self-administered behavioural risk assessment, and re-starting PrEP | 1 year
  In-Depth Interviews will be conducted to collect participant's experience while in the study and tools used during the study.

CONTACTS AND LOCATIONS:
Locations (1):
- Wits RHI Research Centre, Hillbrow, Gauteng, South Africa

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all outcome measures will be made available after study completion.
Supporting Information: Study Protocol, ICF
Access Criteria: A data request from the PI needs to be made before the data can be released

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-10-13): https://cdn.clinicaltrials.gov/large-docs/56/NCT06030856/Prot_SAP_000.pdf
  • Informed Consent Form (2022-12-19): https://cdn.clinicaltrials.gov/large-docs/56/NCT06030856/ICF_001.pdf